CLINICAL TRIAL: NCT02889003
Title: Combination Study of Pioglitazone and Tyrosine Kinase Inhibitors (TKIs) in Chronic Myeloid Leukemia Patients After Failure of a First TKIs Discontinuation Attempt in Order to Prepare a New Stop
Brief Title: Second STOP After Pioglitazone Priming in CML Patients
Acronym: PIO2STOP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Versailles Hospital (Other)
Collaborators: Pr Philippe ROUSSELOT (Unknown)
Responsible Party: Principal Investigator, Dr Noémie DE GUNZBURG, Investigator coordinator, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P16/05_PIO2STOP
Record Dates: First submitted 2016-08-19; First posted 2016-09-05 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Chronic Myeloid Leukemia (CML)
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CML patients following molecular response loss (Experimental)
  Interventions: Drug: Pioglitazone + TKI

INTERVENTIONS:
Drug: Pioglitazone + TKI

SUMMARY:
Single-center study, prospective, phase II trial.

The study objectives are :

* To assess safety and pharmacokinetics of the combination of PIO and TKI in CML subjects who experience a loss of MMR following a first TKI discontinuation.
* To assess survival without loss of MMR over a 12 months period following a second TKI discontinuation in subjects who achieve or maintain < MR4.5 with the combination PIO and TKI administered for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. CML in any phase. patient in MR4
2. Loss of MMR following a first or subsequent TKI discontinuation trial.
3. Patient prior treated with imatinib, dasatinib, nilotinib, or bosutinib
4. Age >18 years.
5. Serum bilirubin <1.5 x upper limit of normal values.
6. AST (SGOT)/ALT (SGPT) <2.5x upper limit of normal values.
7. Females of child bearing potential must agree to abstain from sexual activity or to use a medically approved contraceptive measure/regimen during and for 3 months after the treatment period. Women of child bearing potential must have a negative urine pregnancy test at the time of enrollment. Acceptable methods of birth control include oral contraceptive, intrauterine device, transdermal/implanted or injected contraceptives and abstinence.
8. Males must agree to abstain from sexual activity or agree to utilize a medically-approved contraception method during and for 3 months after the treatment period.
9. Signed informed consent.
10. Be able and willing to comply with study visits and procedures

Exclusion Criteria:

1. Known loss of CCyR by marrow cytogenetic or blood FISH for BCR-ABL1.
2. Loss of CHR.
3. Participation in another clinical trial with any investigative drug within 30 days prior to study enrolment.
4. Prior allogeneic hematopoietic stem cell transplantation.
5. Patient requiring anti-diabetic medications to manage hyperglycemia.
6. Cardiovascular disease: history of congestive heart failure, myocardial infarction within the 6 months of study entry, symptomatic cardiac arrhythmia requiring treatment.
7. Hepatic insufficiency
8. History of bladder cancer.
9. Diagnosed hematuria.
10. Known osteoporosis with curative therapy (prophylactic therapy is not an exclusion criteria)
11. Known history of macular edema.
12. Known history of ABL1-domain mutation associated with resistance to the discontinued TKI.
13. Known allergy to PIO.
14. Pregnant or breastfeeding.
15. Use of TZD within 28 days prior to enrollment.
16. Significant gastrointestinal condition that could potentially impair the absorption or disposition of the drug.
17. Uncontrolled peripheral edema (2+ or more) of any etiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 24 months after inclusion
Treatment free survival after pioglitazone and tyrosine kinase inhibitor discontinuation. | Up to 24 months after inclusion

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre Hospitalier de Versailles, Le Chesnay
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU de Nantes, Nantes
  - CHU de Rennes, Rennes

IPD SHARING:
Plan to Share IPD: Yes